CLINICAL TRIAL: NCT02537652
Title: Effect of Posture and Fasting State on Central and Peripheral Blood Pressure in Patients With Stroke
Brief Title: Central and Peripheral Blood Pressure in Stroke
Status: Completed | Type: Observational
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Collaborators: University of Winchester (Other)
Responsible Party: Sponsor
Other Study IDs: 184563
Record Dates: First submitted 2015-08-25; First posted 2015-09-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Stroke, Acute; Blood Pressure
Keywords: Central blood pressure; Transient ischaemic attack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Major Stroke: Patients diagnosed with major stroke who will undergo blood pressure assessment
  Interventions: Other: Blood pressure assessment
- Minor stroke: Patients diagnosed with minor stroke who will undergo blood pressure assessment
  Interventions: Other: Blood pressure assessment

INTERVENTIONS:
Other: Blood pressure assessment — Participants will undertake an overnight fast prior to each assessment (only water is allowed to be consumed prior to the assessment). Participants will take their medication the morning of each assessment in accordance with the normal pharmacological management procedures which are used on the acute stroke ward at the Royal Hampshire County Hospital. Following this, participants will rest supine (on an electrically operated bed) for a minimum of 15 minutes. Oscillometric pressure waveforms (using the SphygmoCor XCEL), recorded on the left upper arm, will assess haemodynamic parameters including central and peripheral blood pressure, pulse pressure, and augmentation index (fasted, supine condition).

SUMMARY:
Individuals who experience a stroke or transient ischaemic attack (TIA) are at heightened risk of subsequent vascular events, including heart attacks and secondary stroke/TIA. Blood pressure control is considered the most important contributor to positive health outcomes in stroke patients. The measurement of central blood pressure (cSBP) (the blood pressure which is being exerted at the heart), may provide clinicians with important diagnostic and prognostic information over and above that typically obtained from a peripheral blood pressure measure (the blood pressure in the arm). Central blood pressures may be better than traditional peripheral blood pressure measures as: i) peripheral blood pressure may not accurately reflect the effects of peak arterial blood pressure on centrally located organs, ii) central blood pressures may be 50 % superior to peripheral blood pressures when predicting cardiovascular events, and iii) information pertaining to central blood pressures may be more effective in the management of hypertension. While the validity of oscillometric devices which measure central blood pressures has been demonstrated, further study is required to determine precision under normal clinical operating conditions (i.e., reflective of the Hospital/GP practice setting). As such, this study will assess central and peripheral blood pressures of stroke patients when fasted and nonfasted, and when seated and supine. The study is interested in identifying the effect of the above parameters (fasted vs. unfasted, seated vs. supine) on central and peripheral blood pressures in stroke patients.

Participants will take part in three separate assessment sessions, on three separate days, with a minimum 24 hour recovery between each session. Each assessment is expected to last 90 minutes, with a minimum of eight blood pressures being taken from the left upper arm. As such, participants will be asked to give up 4.5 hours of their time to the study. During each assessment participants will be tested in a fasted and non-fasted state, and in a supine (lying) and seated position. All assessments will take place between 7 and 10am and will be undertaken following written informed consent.

DETAILED DESCRIPTION:
Stroke is a leading cause of death worldwide, and is a prominent cause of chronic disability, causing significant physical, cognitive and social impairment. In the United Kingdom, there are 150,000 strokes each year, with ~900,000 people living with the debilitating effects of stroke.Individuals who experience a stroke or transient ischaemic attack (TIA; minor stroke) are at heightened risk of experiencing vascular events in the future, such as myocardial infarction, stroke and secondary TIAs, and death. Of all the measures of interest, greater blood pressure control is the most important contributor to positive health outcomes in stroke patients. However, clinical practice, and research to date concentrate on the assessment of peripheral blood pressure assessments (the blood pressure as identified from the arm). The measurement of central haemodynamic parameters, including central systolic blood pressure (cSBP) and arterial wave reflection (i.e., augmentation index, AIx), hold the potential to provide clinicians with important diagnostic and prognostic information beyond that provided by traditional peripheral blood pressure readings. The assessment of central blood pressure is important as it reflects the stress and loading on the left ventricle and coronary arteries. Considering the marked differences in pulse pressure between the central aorta and peripheral limbs, peripheral blood pressure may not accurately reflect the effects of peak arterial blood pressure on centrally located organs. Previous research has demonstrated central blood pressures to be 50 % superior to peripheral blood pressures when predicting cardiovascular events, while in comparison to peripheral blood pressure, central blood pressure may improve the management of hypertension. Owing to recent technological advances, central haemodynamic parameters can be obtained quickly and noninvasively using an automated blood pressure cuff (oscillometer).While the validity of these devices which measure central haemodynamic parameters has been demonstrated, further study is required to determine measurement precision (reliability) under normal clinical operating conditions (i.e. , in the hospital or general practioner setting). As such, this study will assess the influence of fasting status (fasted vs. nonfasted) and posture (seated vs. supine) on central and peripheral blood pressure measures in patients diagnosed with stroke. The study will determine whether these parameters can be reliably assessed and whether stroke severity (major stroke, minor stroke, TIA) influences the reported results.

Design and setting:

This study is a single centre observational study. All stroke/TIA patients will be recruited from the Royal Hampshire County Hospital within the Hampshire Hospital NHS Foundation Trust (HHFT).

Patients will be recruited from the inpatient and outpatient setting. For patients diagnosed with a major or minor stroke and who have not been discharged from the hospital, recruitment will take place on the acute stroke ward at the hospital. For these patients, all assessments will also be undertaken within the hospital as patients will be based in the acute stroke ward. For those patients identified with minor stroke or TIA within the emergency department or outpatient setting (i.e., stroke clinics), and who not be staying in the acute stroke ward, will be recruited from these settings. All assessments with these patients will take place in the Physiology Laboratory at the University of Winchester. Written informed consent will be obtained from all participants.

All stroke (minor and major) patients will be assessed using the National Institute of Health Stroke Severity Scale (NIHSS). All patients with suspected TIA with be assessed with the ABCD2. Participants will comply with pharmacological treatment as recommended.

Participants will take part in three separate assessment sessions, on three separate days, with a minimum 24 hour recovery between each session. Before each assessment participants will undertake an overnight fast (only water is allowed to be consumed prior to the assessment). Participants will take their medication the morning of each assessment in accordance with the normal pharmacological management procedures which are used on the acute stroke ward at the Royal Hampshire County Hospital. Following this, participants will rest supine for a minimum of 15 minutes. Oscillometric pressure waveforms (using the SphygmoCor XCEL), recorded on the left upper arm, will assess haemodynamic parameters including central and peripheral blood pressure, pulse pressure, and augmentation index. Two measurements will be taken with a three-minute interval. If peripheral blood pressure is > 5 mmHg or augmentation index is > 4 %, a third measure will be taken. Following this, participants will be moved to a seated position and remain rested for a further 15 minutes. Identical procedures to those outlined above will then be used to assess central and peripheral blood pressure responses. Thereafter, patients will consume their normal breakfast. However, caffeine cannot be consumed during this time. Thirty-minutes after food consumption participants will undertake identical procedures as those outlined above in both a non-fasted-supine and non-fasted-seated conditions.

Identical procedures to those outlined in the first assessment session will be used to assess central and peripheral blood pressure measures during the second and third assessment day.

Oscillometric pressure waveforms will be recorded on the left upper arm using the SphygmoCor XCEL device during all assessments, following standard manufacturer guidelines. Each measurement cycle lasts approximately 60 sec, consisting of a brachial blood pressure recording and then a 10 sec sub-systolic recording. A corresponding aortic pressure waveform will then be generated using a validated transfer function, from which central systolic, diastolic, pulse pressure (cSBP, cDBP, cPP), augmentation pressure (AP), and augmentation index (AIx) will be derived. The AP is defined as cSBP minus the pressure at the inflection point, whereby the inflection point is the merging of the forward and reflected waves. The AIx is defined as the AP expressed as a percentage of cPP. AIx is influenced by heart rate, and thus an index corrected for a heart rate at 75 beats per minute (AIx@75) will also be calculated.

Central and peripheral blood pressures will be assessed in the following four conditions during each of the three assessment sessions: i) fasted, supine, ii) fasted, seated, iii) non-fasted supine, and iv) non-fasted seated. During each of the above conditions two measurements will be taken, separated by a three-minute interval. If blood pressure differ by > 5mmHG a third recording will be taken and the closest recordings will be averaged. Each of the above conditions will be undertaken following a minimum 15 minutes quite rest.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with major stroke, minor stroke or TIA by a member of the clinical team.
* Reside within the locality of the Hampshire Hospital's Foundation Trust
* Patients are to be assessed within 8 weeks of their initial stroke/TIA diagnosis.
* Do not meet exclusion criteria

Exclusion Criteria:

* end of life stroke patients;
* Unstable cardiac conditions
* oxygen dependence
* significant dementia; patients lacking capacity to consent to participate in study
* unable to swallow
* Patient is diagnosed with major stroke, minor stroke or TIA more than 8 weeks prior to an assessment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a major stroke, minor stroke or TIA by a stroke consultant at a local hospital will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Central blood pressure | 10 months
  Central blood pressures will be assessed on three separate days in both a seated and supine posture when fasted and unfasted.

SECONDARY OUTCOMES:
Peripheral blood pressure | 10 months
  Peripheral blood pressures will be assessed on three separate days in both a seated and supine posture when fasted and unfasted.
Augmentation index | 10 months
  Augmentation index will be assessed on three separate days in both a seated and supine posture when fasted and unfasted. Augmentation index is a parameter obtained during the central and peripheral blood pressure assessment (it is not a separate stand alone measure).
  The augmentation index is a ratio calculated from the blood pressure waveform, it is a measure of wave reflection and arterial stiffness.
Pulse pressure | 10 months
  Pulse pressure will be assessed on three separate days in both a seated and supine posture when fasted and unfasted.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mitchelmore, MSc, Principal Investigator — University of Winchester
Locations (2):
- United Kingdom (2):
  - University of Winchester, Winchester, Hampshire
  - Acute Stroke Ward, Winchester, Hampshire

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be anonymised before it is shared outside the clinical study team

REFERENCES:
- [Derived] Mitchelmore A, Stoner L, Lambrick D, Sykes L, Eglinton C, Jobson S, Faulkner J. Oscillometric central blood pressure and central systolic loading in stroke patients: Short-term reproducibility and effects of posture and fasting state. PLoS One. 2018 Nov 1;13(11):e0206329. doi: 10.1371/journal.pone.0206329. eCollection 2018. PMID 30383781